CLINICAL TRIAL: NCT00196911
Title: Randomized, Multicenter, Prospective, Parallel-Group Study of the Effect of Deep Brain Stimulation (Subthalamic Nucleus) on Quality of Life and Motor Complications in Patients With Advanced Parkinson's Disease Compared With Best Medical Treatment
Brief Title: STN-Stimulation Versus Best Medical Treatment in Advanced PD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: German Parkinson Study Group (GPS) (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A 125/00; Grant 01 GI 0201/01 GI 0401
Record Dates: First submitted 2005-09-11; First posted 2005-09-20 (Estimated); Last update posted 2006-11-30 (Estimated); Status verified 2005-09

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

INTERVENTIONS:
Procedure: Implantation of stimulation electrodes in the STN

SUMMARY:
Assessment of the therapeutic effect of deep brain stimulation of the subthalamic nucleus compared with drug treatment alone in patients with advanced Parkinson's disease.

DETAILED DESCRIPTION:
Patients are randomized either to medical treatment or subthalamic stimulation. The observation period was 6 months. The primary outcome criterium: PDQ-39 and UPDRS III.

ELIGIBILITY:
Inclusion Criteria:

advanced Parkinson's disease with UPDRS III score >29/104 or Dyskinesia score > 2 or tremor >2

Exclusion Criteria:

age>75 years depression psychosis surgical contraindications

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156
Dates: Start 2001-01; Study Completion 2005-01

PRIMARY OUTCOMES:
Quality of life
Motor Score in the OFF (UPDRS III)

CONTACTS AND LOCATIONS:
Overall Officials: Guenther Deuschl, Prof., Principal Investigator — Department of Neurology, Christian-Albrechts University
Locations (6):
- Germany (6):
  - Neurologische Klinik der Charité, Augustenburgerplatz 1, Berlin
  - Neurologische Klinik der Universität, Gleuelerstr. 50, Cologne
  - Neurologische Klinik der Universität, Moorenstr. 5, Düsseldorf
  - Neurologische Klinik der Universität, Neuenheimerfeld 400, Heidelberg
  - Department of Neurology, Schittenhelmstr. 10, Kiel
  - Neurologische Klinik der Universität, München

REFERENCES:
- [Result] Deuschl G, Schade-Brittinger C, Krack P, Volkmann J, Schafer H, Botzel K, Daniels C, Deutschlander A, Dillmann U, Eisner W, Gruber D, Hamel W, Herzog J, Hilker R, Klebe S, Kloss M, Koy J, Krause M, Kupsch A, Lorenz D, Lorenzl S, Mehdorn HM, Moringlane JR, Oertel W, Pinsker MO, Reichmann H, Reuss A, Schneider GH, Schnitzler A, Steude U, Sturm V, Timmermann L, Tronnier V, Trottenberg T, Wojtecki L, Wolf E, Poewe W, Voges J; German Parkinson Study Group, Neurostimulation Section. A randomized trial of deep-brain stimulation for Parkinson's disease. N Engl J Med. 2006 Aug 31;355(9):896-908. doi: 10.1056/NEJMoa060281. PMID 16943402
- [Derived] Daniels C, Krack P, Volkmann J, Raethjen J, Pinsker MO, Kloss M, Tronnier V, Schnitzler A, Wojtecki L, Botzel K, Danek A, Hilker R, Sturm V, Kupsch A, Karner E, Deuschl G, Witt K. Is improvement in the quality of life after subthalamic nucleus stimulation in Parkinson's disease predictable? Mov Disord. 2011 Dec;26(14):2516-21. doi: 10.1002/mds.23907. Epub 2011 Aug 25. PMID 22170276
- [Derived] Witt K, Daniels C, Krack P, Volkmann J, Pinsker MO, Kloss M, Tronnier V, Schnitzler A, Wojtecki L, Botzel K, Danek A, Hilker R, Sturm V, Kupsch A, Karner E, Deuschl G. Negative impact of borderline global cognitive scores on quality of life after subthalamic nucleus stimulation in Parkinson's disease. J Neurol Sci. 2011 Nov 15;310(1-2):261-6. doi: 10.1016/j.jns.2011.06.028. Epub 2011 Jul 5. PMID 21733529
- [Derived] Daniels C, Krack P, Volkmann J, Pinsker MO, Krause M, Tronnier V, Kloss M, Schnitzler A, Wojtecki L, Botzel K, Danek A, Hilker R, Sturm V, Kupsch A, Karner E, Deuschl G, Witt K. Risk factors for executive dysfunction after subthalamic nucleus stimulation in Parkinson's disease. Mov Disord. 2010 Aug 15;25(11):1583-9. doi: 10.1002/mds.23078. PMID 20589868
- [Derived] Witt K, Daniels C, Reiff J, Krack P, Volkmann J, Pinsker MO, Krause M, Tronnier V, Kloss M, Schnitzler A, Wojtecki L, Botzel K, Danek A, Hilker R, Sturm V, Kupsch A, Karner E, Deuschl G. Neuropsychological and psychiatric changes after deep brain stimulation for Parkinson's disease: a randomised, multicentre study. Lancet Neurol. 2008 Jul;7(7):605-14. doi: 10.1016/S1474-4422(08)70114-5. Epub 2008 Jun 4. PMID 18538636
- See also: German Research Collaboration, funded by the German Ministery of Research — http://www.kompetenznetz-parkinson.de/
- See also: Homepage Coordination Center for Clinical Studies to STN Study, Language: German — http://www.kks-mr.de